CLINICAL TRIAL: NCT01459484
Title: ABCB1/P-glycoprotein Expression as Biologic Stratification Factor for Patients With Non Metastatic Osteosarcoma - Prospective Study (ISG/OS-2)
Brief Title: ABCB1/P-glycoprotein Expression as Biologic Stratification Factor for Patients With Non Metastatic Osteosarcoma
Acronym: ISG/OS-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISG/OS-2; 2011-001659-36 (EudraCT Number)
Record Dates: First submitted 2011-10-19; First posted 2011-10-25 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Osteosarcoma
Keywords: Non metastatic extremities high grade osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Methotrexate; Cisplatin; Doxorubicin; Ifosfamide; mifamurtide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mifamurtide arm (Experimental): Chemotherapy for patients who over express ABCB1/P-glycoprotein (methotrexate, cisplatinum, doxorubicine, ifosfamide + mifamurtide)
  Interventions: Drug: Mifamurtide arm
- 3 drugs arm (Other): High grade osteosarcoma treatment for patients who do not over express ABCB1/P-glycoprotein
  Interventions: Other: 3 drugs arm

INTERVENTIONS:
Drug: Mifamurtide arm — PRE SUGERY TREATMENT:
  Methotrexate: 12g/m2 (3 cycles) Cisplatinum: 120mg/m2 (3 cycles) Doxorubicin: ADM 75mg/m2 (3 cycles)
  POST SURGERY TREATMENT for good responder patients with positive P-GLYCOPROTEIN
  Methotrexate 12g/m2 (10 Cycles) Cisplatinum 120mg/m2; Doxorubicin 90mg/m2 MEPACT 2 mg/m2 twice a week for the first 3 months the weekly for the next 6 months (total lenght treatment 44 weeks)
  POST SURGERY TREATMENT for poor responder patients with positive P-GLYCOPROTEIN
  Methotrexate 12g/m2; Cisplatinum 120mg/m2; Doxorubicin 90mg/m2 ifosfamide 15g/m2 MEPACT 2 mg/m2 twice a week for the first 3 months the weekly for the next 6 months (total lenght treatment 44 weeks)
  All the product are used as commercial formulation
  Other Names: Methotrexate; Cisplatinum; doxorubicin; ifosfamide; mifamurtide
  Arms: Mifamurtide arm
Other: 3 drugs arm — High grade osteosarcoma who do not over express ABCB1/P-glycoprotein will be treated with a standard 3-drugs regimen
  PRE-SUGERY TREATMENT:
  Methotrexate: 12g/m2 (3 cycles) Cisplatinum: 120mg/m2 (3 cycles) Doxorubicin: ADM 75mg/m2 (3 cycles)
  POST SURGERY TREATMENT:
  Methotrexate 12g/m2 (10 cycles) Cisplatinum 120mg/m2; Doxorubicin 90mg/m2
  Total lenght 34 weeks
  All the product are used as commercial formulation
  Other Names: methotrexate; cisplatin; doxorubicine
  Arms: 3 drugs arm

SUMMARY:
This is a phase II multicentre, uncontrolled trial including patients ≤ 40 years with non-metastatic extremity high-grade osteosarcoma stratified according to P-glicoprotein expression

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the impact on event-free survival (EFS) of a multi-drug chemotherapy approach and mifamurtide treatment in patients with non-metastatic osteosarcoma of the extremities according to the expression of ABCB1/P-glycoprotein

ELIGIBILITY:
Inclusion Criteria:

* Histology confirmed diagnosis of extremities high grade osteosarcoma
* Age ≤ 40 years
* Localized disease or presence of skip metastasis
* Hepatic, renal and bone marrow normal function
* LVEF > 50%
* No previous surgery and/ or chemotheraputic osteosarcoma treatments,
* No more than 4 weeks interval between histological diagnosis and start of chemotherapy
* Informed consent to the study participation obtained.

Exclusion Criteria:

* Presence of metastases other than skip metastases
* Periosteal Osteosarcoma, parostal osteosarcoma, secondary osteosarcoma,
* Medical contra-indication to the drugs foreseen in the protocol,
* Subject is pregnant or breast feeding
* Mental or social conditions that can compromise a correct adherence to the protocol and its procedures

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 225 (Actual)
Dates: Start 2011-06-23 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Events free survival | After 5 years from the time to first day of chemotherapy for all patients and from the date of surgery for the Pgp overexpression patients stratified according to tumor necrosis (Good Responders and Poor Responders).
  Onset of any event. An event is the defined as disease recurrence (local or distant), death for disease or any other cause, onset of secondary tumors or the last follow-up examination

SECONDARY OUTCOMES:
Overall Survival | After 5 years from the time to first day of chemotherapy for all patients and from the date of surgery for the Pgp overexpression patients stratified according to tumor necrosis (Good Responders and Poor Responders).
  Time elapsed for the diagnosis to the death for any cause or to the last follow-up examination.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Palmerini, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (11):
- Italy (11):
  - I.R.C.C. - Unit of Medical Oncology, Candiolo, Torino
  - Presidio Sanitario Gradenigo, Torino, TO
  - IRCCS Istituto ortopedico Rizzoli, Bologna
  - A.O. Universitaria Meyer, Florence
  - Istituto Giannina Gaslini, Genova
  - FONDAZIONE IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Nazionale Tumori "Fondazione G. Pascale", Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Istituti Fisioterapici Ospitalieri di Roma, Roma
  - Ospedale Pediatrico Bambin Gesu', Roma
  - Ospedale Infantile Regina Margherita - Unit of Paediatric Oncoematology, Torino

REFERENCES:
- [Background] Serra M, Pasello M, Manara MC, Scotlandi K, Ferrari S, Bertoni F, Mercuri M, Alvegard TA, Picci P, Bacci G, Smeland S. May P-glycoprotein status be used to stratify high-grade osteosarcoma patients? Results from the Italian/Scandinavian Sarcoma Group 1 treatment protocol. Int J Oncol. 2006 Dec;29(6):1459-68. PMID 17088985
- [Derived] Palmerini E, Meazza C, Tamburini A, Marquez-Vega C, Bisogno G, Fagioli F, Ferraresi V, Milano GM, Coccoli L, Rubio-San-Simon A, Gallego O, Llinares Riestra ME, Manzitti C, Mora J, Vaz-Salgado MA, Luksch R, Mata C, Pierini M, Carretta E, Cesari M, Paioli A, Marrari A, Scotlandi K, Serra M, Asaftei SD, Gambarotti M, Picci P, Ferrari S, Valverde C, Ibrahim T, Broto JM. Is There a Role for Mifamurtide in Nonmetastatic High-Grade Osteosarcoma? Results From the Italian Sarcoma Group (ISG/OS-2) and Spanish Sarcoma Group (GEIS-33) Trials. J Clin Oncol. 2025 Oct;43(28):3113-3122. doi: 10.1200/JCO-25-00210. Epub 2025 Aug 18. PMID 40825172
- [Derived] Palmerini E, Meazza C, Tamburini A, Bisogno G, Ferraresi V, Asaftei SD, Milano GM, Coccoli L, Manzitti C, Luksch R, Serra M, Gambarotti M, Donati DM, Scotlandi K, Bertulli R, Favre C, Longhi A, Abate ME, Perrotta S, Mascarin M, D'Angelo P, Cesari M, Staals EL, Marchesi E, Carretta E, Ibrahim T, Casali PG, Picci P, Fagioli F, Ferrari S. Phase 2 study for nonmetastatic extremity high-grade osteosarcoma in pediatric and adolescent and young adult patients with a risk-adapted strategy based on ABCB1/P-glycoprotein expression: An Italian Sarcoma Group trial (ISG/OS-2). Cancer. 2022 May 15;128(10):1958-1966. doi: 10.1002/cncr.34131. Epub 2022 Feb 24. PMID 35201621
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903